CLINICAL TRIAL: NCT02314949
Title: A Multifactorial Immunomodulatory Protocol -Promoting T-regulatory Cells- Prolongs Graft and Patient Survival After Intestinal Transplantation
Brief Title: Leuven Tolerogenic Protocol for Intestinal Transplantation
Acronym: LP
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: LPs56862
Record Dates: First submitted 2014-11-26; First posted 2014-12-11 (Estimated); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Organ Transplantation; Intestine
Keywords: T-regulatory cells; Tolerogenic protocol; immunomodulation
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- intestinal transplantation: all performed intestinal transplants underwent the same Leuven intestinal transplant protocol
  Interventions: Procedure: intestinal transplantation

INTERVENTIONS:
Procedure: intestinal transplantation

SUMMARY:
An immunomodulatory protocol, experimentally-proven to promote T-regulatory dependent graft protective mechanisms was applied in a clinical cohort of 13 intestinal transplant recipients to activate - in a protolerogenic environment - T-regulatory cells.

This protocol is the standard of care in the investigators intestinal transplant programme since the first intestinal transplant was performed in october 2000.

DETAILED DESCRIPTION:
The LP is a 4-step approach that aims to upregulate T-regulatory cells (T-Regs) by directly stimulating their development and removing stimuli that could suppress them, eventually creating an environment favorable for graft acceptance. This protocol has been based upon preclinical research perormfed in the investigators lab and has been implemented as standard of care since the inception of the clinical programma in 2000. Patients gave informed consent for Donor Specific Blood Transfusion. Ethical approval for collection of additional blood samples was granted by the local ethical committee (s56862).

Step 1. Donor-specific blood transfusion (DSBT). 400 mL of whole blood was collected from the donor at the time of procurement and was transfused systemically in the recipient prior to reperfusion.

Step 2. Avoiding high-dose steroids. After Intestinal Transplantation, only 16 mg of medrol was administered and tapered towards 4 mg in 3 to 6 months post-Tx, similar to the liver Tx protocol.

Step 3. Avoiding high-dose calcineurin inhibitors (tacrolimus). Initial levels of 15 ng/ml were tapered -within 3 to 6 months- to 5 ng/mL or less for liver-containing grafts and 6 to 8 ng/mL for isolated intestinal grafts.

Step 4. Maintaining mucosal integrity and reducing ischemia reperfusion injury, inflammation, and endotoxin translocation. This was obtained by selecting perfect (ischemia-free) donors (<50y, absence of significant hypotension, vasopressor requirement and cardiac arrest); pretreating donors with selective bowel decontamination and glutamine; gentle manipulations of the organs during donor and recipient surgery; aiming for short cold and warm ischemic times (5h and 30' respectively). Bowel decontamination consists of Nilstat, Tobramycine and Colimycine administered by a nasogastric tube and continued posttransplant during three months. Glutamine is supplemented parenterally (Dipeptiven Kabi Fresenius) and enterally (Alitracq) to donors and continued posttransplant.

ELIGIBILITY:
Inclusion Criteria:

* all patients awaiting intestinal transplantation

Exclusion Criteria:

* living donation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent intestinal transplantation
Sampling Method: Non-Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2000-10; Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 10 years
  routine clinical follow-up and Kaplan Meier Analysis

SECONDARY OUTCOMES:
T-regulatory cells CD4+ CD45RA- Foxp3hi | 10 years
  Peripheral blood mononuclear cells (PBMC's) isolation and flow cytometry
rejection | 10 years
  routine endoscopical obtained ileal biopsies analysed for number of apoptotic bodies in the crypt

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Ceulemans LJ, Braza F, Monbaliu D, Jochmans I, De Hertogh G, Du Plessis J, Emonds MP, Kitade H, Kawai M, Li Y, Zhao X, Koshiba T, Sprangers B, Brouard S, Waer M, Pirenne J. The Leuven Immunomodulatory Protocol Promotes T-Regulatory Cells and Substantially Prolongs Survival After First Intestinal Transplantation. Am J Transplant. 2016 Oct;16(10):2973-2985. doi: 10.1111/ajt.13815. Epub 2016 May 12. PMID 27037650